CLINICAL TRIAL: NCT04625530
Title: Perioperative Management With Ferric Carboxymaltose and Tranexamic Acid to Reduce Transfusion Rate in Gynaecological Carcinoma Surgery: a Single-blind, Mono-centre, Randomized Trial
Brief Title: Perioperative Management in Gynaecological Carcinoma Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Issue with grant transfer upon sponsor relocation
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01194; sp20Amstad
Record Dates: First submitted 2020-11-04; First posted 2020-11-12 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Gynaecological Carcinoma
Keywords: ferric carboxymaltose; tranexamic acid; RBC transfusion
MeSH Terms: interventions — ferric carboxymaltose; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be blinded to participants and statistician conducting the data analysis. The physicians and nurses who will perform this infusion will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ferric carboxymaltose (Experimental): ferric carboxymaltose 20 mg/kg (with a maximum dose of 1000 mg ferric carboxymaltose in a single Infusion) (Ferinject® 1000 mg/20 ml) will be administered between day -27 and day -7.
  Interventions: Drug: ferric carboxymaltose
- tranexamic acid (Experimental): tranexamic acid 10mg/kg (Tranexam OrPha 1000 mg/10 ml, OrPha Swiss GmbH, Küsnacht, Switzerland) will be administered 15 -30 minutes prior to surgery followed by infusion of tranexamic acid through syringe pump (1 mg/kg/h) till 4 h postoperatively
  Interventions: Drug: tranexamic acid
- ferric carboxymaltose and tranexamic acid (Experimental): ferric carboxymaltose (Ferinject® 1000 mg/20 ml) between day -27 and day
  -7 and tranexamic acid (Tranexam OrPha 1000 mg/10 ml) 15-30 minutes prior to surgery followed by Infusion of tranexamic acid through syringe pump (1 mg/kg/h) till 4 h postoperatively will be administered.
  Interventions: Drug: ferric carboxymaltose and tranexamic acid
- no treatment accordingly "current standard of care" (No Intervention): no treatment accordingly "current standard of care" will be given

INTERVENTIONS:
Drug: ferric carboxymaltose — Ferric carboxymaltose 20 mg/kg (with a maximum dose of 1000 mg ferric carboxymaltose in a single Infusion) (Ferinject® 1000 mg/20ml, Vifor (International) AG, St. Gallen, Switzerland) will be diluted in 250 ml of 0.9% m/V sodium chloride solution and administered over 15 minutes intravenously between day -27 and day -7. The colour of ferric carboxymaltose is dark brown. A single Ferinject administration should not exceed 20 mg iron/kg body weight.
  Arms: ferric carboxymaltose
Drug: tranexamic acid — Tranexamic acid 10mg/kg (Tranexam OrPha 1000 mg/10 ml, OrPha Swiss GmbH, Küsnacht, Switzerland) will be administered 15 -30 minutes prior to surgery followed by infusion of tranexamic acid through syringe pump (1 mg/kg/h) till 4 h postoperatively. The colour of the medicament is transparent.
  Arms: tranexamic acid
Drug: ferric carboxymaltose and tranexamic acid — Ferric carboxymaltose (Ferinject® 1000 mg/20 ml) will be administered between day -27 and day -7 and tranexamic acid (Tranexam OrPha 1000 mg/10 ml) 15-30 minutes prior to surgery followed by infusion of tranexamic acid through syringe pump (1 mg/kg/h) till 4 h postoperatively.
  Arms: ferric carboxymaltose and tranexamic acid

SUMMARY:
This study is to determine the effect of perioperative treatment with intravenous iron and tranexamic acid on the reduction of intraoperative and postoperative RBC transfusions in gynaecological carcinoma patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Radical abdominal surgery often leads to intraoperative bleeding frequently exceeding 1000 ml and approximately 50% of women undergoing this surgery require blood transfusion. Perioperative blood transfusions have been shown to increase of length of stay, surgical complications, postoperative morbidity and mortality. There are a few data on the reduction in red blood cell count (RBC) transfusions using perioperative management with intravenous iron and tranexamic acid in women with gynaecological carcinoma surgery. This study is to determine the effect of perioperative treatment with intravenous iron and tranexamic acid on the reduction of intraoperative and postoperative RBC transfusions in gynaecological carcinoma patients undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* informed consent as documented by signature
* women with gynaecological carcinoma surgery with hemoglobin level between 90-120 g/I and serum ferritin < 100 µg/I (or ferritin index < 3.19) at recruitment
* pregnancy test negative in women younger than 50 years

Exclusion Criteria:

* known hypersensitivity or allergy to ferric carboxymaltose or tranexamic acid
* history or present laboratory signs of bleeding disorders, coagulopathy or thromboembolic events
* history of myocardial infarction within the last year, present unstable angina or severe coronary disease
* increased plasma creatinine levels above 250 µmol/I
* inability to follow the procedures of the study (language problems, severe psychiatric or mental disorders)
* iron overload
* current administration of intravenous iron or previous intravenous iron therapy or blood transfusion within three months
* date of scheduled surgery is outside 28 days after the date of recruitment
* other clinically significant concomitant disease states (e.g., hepatic dysfunction, cardiovascular disease, etc.)
* participation in another study with investigational drug within the 30 days
* enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
number of all perioperative (intraoperative and postoperative) administered RBC transfusions | day of surgery until follow up visit 5 (up to 28 days)
  number of all perioperative (intraoperative and postoperative) administered RBC transfusions (the absolute rate of RBC transfusions)

SECONDARY OUTCOMES:
change in hemoglobin level | day of surgery until follow up visit 5 (up to 28 days)
  change in hemoglobin level (g/dl)
rate of transfused women with gynaecological carcinoma during and/or after surgery | day of surgery until follow up visit 5 (up to 28 days)
  rate of transfused women with gynaecological carcinoma during and/or after surgery
blood loss measured during surgery (ml) | day of surgery
  blood loss measured during surgery (ml)
rate of other blood product transfusions | day of surgery until follow up visit 5 (up to 28 days)
  rate of other blood product transfusions (fresh frozen plasma, autologous whole blood)
requirement of additional local or systematic haemostatic therapy (descriptive) | day of surgery until follow up visit 5 (up to 28 days)
  requirement of additional local or systematic haemostatic therapy (descriptive)
duration of surgery (minutes) | day of surgery
  duration of surgery (minutes)
duration of hospitalisation (days) | from admission to discharge date (up to 56 days)
  duration of hospitalisation (days)
number of postoperative complications | day of surgery until follow up visit 5 (up to 28 days)
  number of postoperative complications: abdominal pain, haemorrhage, reoperation owing to bleeding, wound infection, pulmonary complications, postoperative renal dysfunction, systemic sepsis
postoperative mortality | day of surgery until follow up visit 5 (up to 28 days)
  postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Amstad Bencaiova, Dr. med., Principal Investigator — Department of Obstetrics and Gynaecology, University Hospital Basel
Locations (1):
- Department of Obstetrics and Gynaecology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data generated by our research will be available as soon as possible, wherever legally and ethically possible. The data will be made available upon reasonable request. The deidentified participant data from this study and related documents (study protocol, statistical analysis plan, patient consent form) will be made available upon request. Researchers may request data to repeat the analyses or use the data for secondary analyses (e. g., systematic review and meta-analysis). Changes to this plan will be noted in the Data Availability Statement and updated in the registry record (to comply with ICMJE recommendations).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available upon reasonable request for one month.